CLINICAL TRIAL: NCT05397028
Title: Weight Management for the Remission of Type 2 Diabetes Using a Proprietary Meal Replacement System- Diabetes Remission Study (DRS)
Acronym: DRS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient number of subjects
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Warren Peters, MD, MPH, Director, Center for Health Promotion, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5200281
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
Keywords: obesity; Diabetes, Type 2; meal replacement; diabetes remission
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Replace meals with a plant-based meal replacement and self-prepared Meditteranean meals for a max 1200 calorie per day. Enroll in a 12 week intensive lifestyle intervention program.
  Interventions: Dietary Supplement: Meal replacement system; Behavioral: Intensive lifestyle Intervention
- Standard of Care Group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Meal replacement system — Participants will replace meals with a meal replacement system to assess the efficacy of weight loss leading to remission of diabetes (optimal A1C levels).
  Arms: Intervention Group
Behavioral: Intensive lifestyle Intervention — Participants will sign up with a virtual health program which they will interact with.
  Arms: Intervention Group

SUMMARY:
A three month meal replacement dietary system which combines meal replacements and self-prepared meals which hypothetically will result in Diabetes remission in >30% of intervention subjects

To assess the efficacy of which patients with Type 2 Diabetes (non insulin dependent) can be brought into a optimal A1C remission state without the use of medications by achieving clinically significant weight loss (>20-30 pounds) using a proprietary meal replacement system associated with a 3-month intensive lifestyle program.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Ages 25-65
* Have been diagnosed with non-insulin dependent diabetes for less than five years
* Are taking at least one oral agents for diabetes
* English speaking

Exclusion Criteria:

* Individuals currently being treated for cancer
* Had a myocardial infarction in the previous 3 months
* Have uncontrolled persistent hypertension - diastolic >90 systolic >160
* Individuals with established eating disorder diagnoses
* Individuals who have recent weight loss attempt in the last 3 months with > 5-pound loss
* Use of anti-obesity medications in the last three months
* Individuals who have had bariatric surgery
* Individuals taking medications that are known to cause weight gain including but not limited to insulin, steroids, haloperidol clozapine, risperidone, olanzapine, amitriptyline imipramine, paroxetine, and lithium
* Individuals who are pregnant or planning to become pregnant in the next 6 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of plant-based meal replacement system on A1-C levels | Change between baseline and six month visit.
  Blood draw to measure the effect of the diet on the A1-C level. Normal A1C is at or below 5.7%. Prediabetes levels range between 5.8%-6.4%. Diabetes is at or above 6.5%.

SECONDARY OUTCOMES:
Efficacy of plant-based meal replacement system on insulin levels | Change between baseline and six month visit.
  Blood draw to measure the effect of the diet on fasting insulin. Insulin levels under the value 10 are considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Peters, MD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No